CLINICAL TRIAL: NCT02910752
Title: Salavge Chemotherapy With Cladribine, Cytarabine and Mitoxantrone Followed by Mobilized Peripheral Stem Cell Infusion From the Original Donor for Relapsed Patients After Allogeneic Stem Cell Transplantation: Phase I/II Study
Brief Title: CLAM Chemotherapy With PBSC Support for Relapsed Patients After Allogeneic Stem Cell Transplantation
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Program, Chief Physician, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allo-HSCT-relapse-2015
Record Dates: First submitted 2016-09-07; First posted 2016-09-22 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLAM|PBSC (Experimental): CLAM chemotherapy with mobilized PBSC infusion: Cladribine 5mg/m2 + cytarabine 1.5g/m2 + mitoxantrone 10mg/m2 from D1 to D5
  Interventions: Drug: CLAM+PBSC

INTERVENTIONS:
Drug: CLAM+PBSC — Cladribine 5mg/m2 + cytarabine 1.5g/m2 + mitoxantrone 10mg/m2 from D1 to D5
  Other Names: CLAMP

SUMMARY:
For acute leukemia patients with early relapse after allogeneic stem cell transplantation, the overall outcome is poor. In this study, we evaluate the treatment outcome and safety of chemotherapy with Cladribine, cytarabine and mitoxantrone followed by peripheral stem cell support from the original donor.

DETAILED DESCRIPTION:
For acute leukemia patients experienced relapse 6 months or less after allogeneic stem cell transplantation, the overall outcome is poor. In this study, we design a treatment protocol aiming to achieve complete remission for this high-risk group of patients with chemotherapy consisting of Cladribine (5mg/m2), cytarabine (1.5g/m2) and mitoxantrone （10mg/m2）for 5 days followed by infusion of mobilized peripheral stem cell from the original donor. For patients who failed to achieved remission,a second cycles will be given. For patients who achieved remission, the post-remission therapy is open depend on patient's intent: consolidation with one more cycle, second allo-HSCT with different donor or continuous DLI.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute leukemia relapsed within 6 months after previous allo-HSCT
* no active GVHD
* mobilized PBSC from the original donor available

Exclusion Criteria:

* ECOG >=3
* liver function/renal function damage (over 2 X upper normal range)
* active infection including CMV and EBV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
complete remission (Bone marrow) | 30 days after treatment
  bone marrow aspiration performed on D30 after treatment. In case of less 5% blast with fully recovery of peripheral blood count is considered as CR. In case of less than 5% blast without fully recovered CBC is considered as CRi

SECONDARY OUTCOMES:
chimerism (bone marrow) | 30 days after treatment
  chiremism analysis of patients bone marrow mononucleared cells at day 30 after treatment
survival | 6 months
  patients remain alive 6 months after enrollment
relapse (bone marrow) | 6 months
  bone marrow relapse within 6 months after treatment
non-relapse mortality | 6 months
  patients died due to any treatment complication or other cause except for disease progression or relapse
GVHD (clinical evaluation and grading) | 6 months
  grade II-IV acute GVHD and cGVHD if presented

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, M.D.,, Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Rui Jin Hospital, Department of Hematology, Shanghai, China

IPD SHARING:
Plan to Share IPD: No